CLINICAL TRIAL: NCT05446220
Title: Twelve-year Follow-up on the Treatment of Obese Pregnant Women (TOP) Study
Acronym: TOP12
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other); Statens Serum Institut (Other); Lund University (Other); University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TOP12
Record Dates: First submitted 2022-07-01; First posted 2022-07-06 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Lifestyle, Healthy; Diet, Healthy; Follow-up; Physical Activity; Body Composition; Gestational Weight Gain
MeSH Terms: conditions — Obesity; Motor Activity; Gestational Weight Gain

STUDY DESIGN:
Intervention Model Description: Follow-up study on healthy lifestyle intervention during pregnancy (randomized controlled trial - TOP study) 12 years after the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diet + physical activity (Experimental): Dietary advise and advise on physical activity monitored by pedometer
  Interventions: Behavioral: Lifestyle intervention
- Physical activity (Experimental): Advise on physical activity monitored by pedometer
  Interventions: Behavioral: Lifestyle intervention
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Lifestyle intervention — Dietary advise and/or advise on physical activity monitored by pedometer
  Arms: Diet + physical activity; Physical activity

SUMMARY:
The participant (both mother and child) in the initial TOP study will be invited to a follow-up study to evaluate the effect of life style intervention during pregnancy on both mother and their offspring 12 years after the intervention. The study will contribute to understanding the transfer of obesity between generations and how to treat as well as prevent obesity.

DETAILED DESCRIPTION:
The initial study (Treatment of Obese Pregnant women (TOP) study) was performed at Hvidovre Hospital, University of Copenhagen in 2009-12 and included 425 pregnant women with pre-gestational BMI ≥ 30kg/m2 in gestational week 11-14. They were randomized 1:1:1 into: 1) a low-calorie Mediterranean-style diet and pedometer assisted physical activity (PA) intervention 2) a pedometer assisted PA intervention alone or 3) no intervention (control). Primary outcome was gestational weight gain (GWG). 389 women completed the study.

The participants (both mother and child in pair) who completed the initial TOP study will be invited to a 3-hour examination now 12 years after the intervention during pregnancy to evaluate the effect of the intervention on both mother and child long term.

ELIGIBILITY:
Inclusion Criteria:

* Participants/mothers in the initial TOP study will be invited with their offspring born following the pregnancy during the initial study to the 12-year follow-up study

Exclusion Criteria:

* There are no exclusion criteria as the potential study population has already been selected at the baseline study in 2009-2012

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 497 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
Body composition | 2 years data collection
  Fatt mass index offspring, DXA scan + BMI mothers

SECONDARY OUTCOMES:
Metabolic and inflammatory markers | 2 years data collection
  Analyses of blood samples
Blood pressure | 2 years data collection
  Standardized sitting measurement of systolic and diastolic blood pressure, average of 3 measures
Glycemic variability | 2 years data collection
  CGM measures
Mental health | 2 years data collection
  Assessed by questionnaires, validated to mother and child respectively
Diet composition | 2 years data collection
  Assessed by FFQ (food frequency questionnaire), validated to mother and child respectively
Level and pattern of physical activity | 2 years data collection
  Assessed by activity tracker worn on the rist for 7 days + IPAQ short (International physical activity questionnaire)
Relative fitness level | 2 years data collection
  Estimated relative fitness level assessed by a submaximal step test (The Danish Step Test)
Epigenetic examinations | 2 years data collection
  Epigenetic examinations
Liver stiffness | 2 years data collection
  FibroScan
Lung function | 2 years data collection
  Spirometry assessing FVC and FEV1
Large artery stiffness | 2 years data collection
  SphygmoCor examination
Eye examination | 2 years data collection
  OPTOS
Sex hormones | 2 years data collection
  Analyses of blood samples, children
Puberty stage | 2 years data collection
  According to the classifications of Marshall and Tanner

CONTACTS AND LOCATIONS:
Overall Officials: Kristina M Renault, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Steno Diabetes Center Copenhagen, Herlev, Denmark